CLINICAL TRIAL: NCT00328198
Title: A Phase II Trial to Evaluate the Efficacy and Safety of Subcutaneously Administered Alemtuzumab (CAMPATH®, MabCampath®) in Patients With Previously Treated B-Cell Chronic Lymphocytic Leukemia
Brief Title: Subcutaneous Alemtuzumab (CAMPATH®, MabCampath®) in Relapsed/Refractory B-Cell Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM203; 2005-005074-69 (EudraCT Number)
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Results first posted 2012-08-10 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-02

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia (B-CLL)
Keywords: CAMPATH; Alemtuzumab; Leukemia; MabCampath; Chronic; Subcutaneous; CLL; C-CLL; Relapsed; Refractory; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Bronchiolitis Obliterans Syndrome; Recurrence | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose escalation (Experimental): Alemtuzumab is administered using escalating doses and alternating injection sites. The dose is escalated as tolerated using 3mg, 10mg, and 30mg administered subcutaneously (SC) (if tolerated).
  Interventions: Biological: Alemtuzumab
- No escalation (Experimental): Alemtuzumab treatment is started immediately at the 30mg dose (with no escalation period), administered subcutaneously at alternating injection sites 3 times per week for up to 18 weeks.
  Interventions: Biological: Alemtuzumab

INTERVENTIONS:
Biological: Alemtuzumab — Alemtuzumab is administered using escalating doses and alternating injection sites. The dose is escalated as tolerated using 3mg, 10mg, and 30mg administered subcutaneously (SC) (if tolerated). When escalation to 30 mg is tolerated, all subsequent doses are administered at 30 mg SC 3 times per week at alternating injection sites for up to 18 weeks.
  Part 1 of the study: The first 20 patients will be randomized to either Arm 1 (dose escalation) or Arm 2 (no escalation). Part 1 of the study has been completed; no additional patients will be enrolled in Part 1. An assigned review panel has reviewed the safety data from Part 1 and determined that all patients will be enrolled and treated under a no escalation schedule for Part 2 of the study.
  Other Names: Campath®, MabCampath®
  Arms: Dose escalation
Biological: Alemtuzumab — Alemtuzumab treatment is started immediately at the 30mg dose (with no escalation period), administered SC at alternating injection sites 3 times per week for up to 18 weeks.
  Part 2 of the study: All patients are currently being enrolled under the no escalation schedule for Part 2 of the study. All patients in Part 2 will be treated with 30mg of alemtuzumab (with no escalation period) administered SC (at alternating injection sites) 3 times per week (e.g., Monday, Wednesday, Friday) for up to 18 weeks. Alemtuzumab is to be administered in a supervised medical setting on an outpatient basis for the first three weeks, after which some study centers may allow a home administration option, with one weekly clinic visit. Under the home administration option, alemtuzumab may be administered by the patient or care giver if the patient meets conditions specified in the protocol guidelines for home administration.
  Other Names: Campath®, MabCampath®
  Arms: No escalation

SUMMARY:
This is a Phase II, open-label, prospective, multicenter study to evaluate the efficacy and safety of subcutaneously administered alemtuzumab (CAMPATH, MabCampath) as therapy for patients with relapsed or refractory B-CLL who have been previously treated.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of B-cell chronic lymphocytic leukemia (B-CLL); according to the National Cancer Institute Working Group (NCI WG) Criteria.
* World Health Organization (WHO) performance status of 0, 1, or 2.
* Life expectancy ≥ 12 weeks.
* Previous therapy with at least one but no more than 5 regimens (single agent or combination regimen). One therapy regimen is defined as consecutive, contiguous cycles of the same drug(s) with no treatment interruptions lasting > 3 months.
* Patient requires treatment for CLL per the following criteria: -Rai stage III or IV; -Rai stage 0-II with at least one of the following - evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia; Massive (i.e. greater than 6 cm below the left costal margin) or progressive splenomegaly; Progressive lymphocytosis with an increase of greater than 50% over a 2-month period or an anticipated doubling time of less than 6 months; Lymphocyte count > 100*10^9/L; B symptoms.
* More than 3 weeks since prior chemotherapy. Patient must have recovered from the acute side effects incurred as a result of previous therapy.
* More than 3 weeks since using investigational agents. Patient must have recovered from the acute side effects incurred as a result of previous therapy.
* Serum creatinine and conjugated (direct) bilirubin less than or equal to 2 times the institutional upper limit of normal (ULN) unless secondary to direct infiltration of the liver with CLL.
* Female patients with childbearing potential must have a negative pregnancy test (serum or urine) within 2 weeks of first dose of study drug(s). All patients must agree to use an effective contraceptive method while on study treatment, if appropriate, and for a minimum of 6 months following study therapy.
* Signed, written informed consent (in the US, includes The Health Insurance Portability and Accountability Act of 1996 (HIPAA) authorization)

Exclusion Criteria:

* Positive Coombs test and evidence of active hemolysis.
* Platelet count less than 50*10^9/L without splenomegaly.
* History of anaphylaxis following exposure to rat or mouse derived CDR-grafted humanized monoclonal antibodies.
* Previously treated with CAMPATH.
* Previous bone marrow transplant.
* Known central nervous system (CNS) involvement with B-CLL
* Active infection, including human immunodeficiency virus (HIV) positive.
* Active second malignancy.
* Recent documented history (within 2 years) of active tuberculosis (TB), current active TB infection, currently receiving anti-tuberculous medication (e.g., INH, rifampin, streptomycin, pyrazinamide, or others).
* Active hepatitis or a history of prior viral hepatitis B or hepatitis C, or positive hepatitis B serologies. Patients with a positive hepatitis B surface antibody (HBsAb) test with a documented history of prior hepatitis B immunization are eligible as long as other criteria are met (i.e. negative tests for: hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) and hepatitis C virus antibody (HCVAb)).
* Other severe, concurrent diseases (e.g., cardiac or pulmonary disease), mental disorders, or major organ malfunction (liver, kidney) that could interfere with the patient ability to participate in the study.
* Pregnant or nursing women.
* Cytomegalovirus (CMV) positive by polymerase chain reaction (PCR) (above the level of detection). A patient that is PCR positive will require treatment to reduce the viral load to a non-detectable level; but such a patient may be considered for study entry once the infection has been treated.
* Medical condition requiring chronic use of oral corticosteroids at a dose higher than physiologic replacement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2006-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (21):
- United States (7):
  - Moores Cancer Center, La Jolla, California
  - Wilshire Oncology Medical Group, La Verne, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - North Mississippi Hematology & Oncology Associates, Ltd., Tupelo, Mississippi
  - Mid Ohio Oncology Hematology, Inc., Columbus, Ohio
  - Joe Arrington Cancer Center, Lubbock, Texas
- Belgium (4):
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
- Czechia (2):
  - University Hospital Brno, Brno
  - University Hospital Hradec Kralove (UH HK), Hradec Králové
- France (3):
  - Hopital Hotel-Dieu, Clermont-Ferrand
  - Hopital Claude Huriez, Lille
  - Hopital Hotel-Dieu, CHU de Nantes-Service d'Hematologie Clinique, Nantes
- Serbia (2):
  - Institute of Hematology, Clinical Centre of Serbia, Belgrade
  - Clinic of Hematology, Clinical Centre Vojvodina Novi Sad, Novi Sad
- United Kingdom (3):
  - Leeds General Infirmary, Leeds
  - Royal Liverpool and Broadgreen Hospitals, Liverpool
  - Nottingham City Hospital, Nottingham

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 109 patients screened and 86 enrolled and treated.
Groups:
- Alemtuzumab 30mg: Participants received a target dose of alemtuzumab 30mg by subcutaneous injection three times a week for up to 18 weeks. Some participants started in the Escalation subpopulation and started at a lower dose and escalated from 3mg to 10 mg to the target 30 mg dose in the first 1-2 weeks.
Period: Treatment
Arm/Group | Alemtuzumab 30mg
Started | 86 (16 participants escalated the dose. 70 participants started at the 30 mg target dose.)
Completed | 48 (Depending upon protocol version, completed treatment was either 12 or 18 weeks in duration.)
Not Completed | 38
Not completed — Adverse Event | 21
Not completed — Death | 1
Not completed — Physician Decision | 5
Not completed — Withdrawal by Subject | 5
Not completed — Evidence of disease progression | 2
Not completed — Non-compliance | 1
Not completed — Confirmed complete response, MRD - | 3
Period: Follow-up
Arm/Group | Alemtuzumab 30mg
Started | 78 (Eight participants did not enter Follow-up)
Completed | 43
Not Completed | 35
Not completed — Lost to Follow-up | 4
Not completed — Death | 31

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab 30mg
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.32 (9.035)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 57
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 82
  Other | 1
Current Rai Stage [Number; unit: participants] — Rai staging is a way to categorize the disease progression of chronic lymphocytic leukemia (CLL); higher stages reflect increasing severity. Data represents the Rai Stage when the participant entered the study.
  Rai Stage 0: Lymphocytosis only, Rai Stage I: Lymphocytosis and lymphadenopathy, Rai Stage II: Lymphocytosis and hepatomegaly +/- splenomegaly, Rai Stage III Lymphocytosis with anemia, Rai Stage IV Lymphocytosis with thrombocytopenia
  participants
    Rai Stage 0 | 7
    Rai Stage I | 10
    Rai Stage II | 22
    Rai Stage III | 7
    Rai Stage IV | 40
Current Binet Stage [Number; unit: participants] — Binet staging is another way to categorize chronic lymphocytic leukemia (CLL). Data represents the Binet Stage when the participant entered the study.
  Stage A CLL is characterized by no anemia or thrombocytopenia and fewer than three areas of lymphoid involvement (Rai stages 0, I, and II).
  Stage B CLL is characterized by no anemia or thrombocytopenia with three or more areas of lymphoid involvement (Rai stages I and II).
  Stage C CLL is characterized by anemia and/or thrombocytopenia regardless of the number of areas of lymphoid enlargement (Rai stages III and IV).
  participants
    Stage A | 20
    Stage B | 22
    Stage C | 44
World Health Organization (WHO) Performance [Number; unit: participants] — The WHO performance status classification categorises patients as:
  0: able to carry out all normal activity without restriction
  1. restricted in strenuous activity but ambulatory and able to carry out light work
  2. ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours
  participants
    0 | 55
    1 | 28
    2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Best Disease Response as Determined by the Independent Response Review Panel (IRRP)
Description: Participants were evaluated by the IRRP according to National Cancer Institute (NCI) 1996 response criteria. The best response observed during the study is summarized. Response categories include Complete Response (CR) with normal physical exam, marrow cells and blood values, Partial Response (PR) with a >= 50% decrease from baseline in lymphocytes, lymphadenopathy and liver or spleen exam, Stable Disease (SD) without significant progression from baseline, or Progressive Disease (PD) with increased size/number of nodes, size of liver or spleen, increase in lymphocytes, aggressive histology.
Time Frame: up to 44 weeks
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Alemtuzumab 30mg
Number analyzed (Participants) | 86
participants
  Overall response (CR+PR) | 37
  Complete response (CR) | 5
  Partial response (PR) | 32
  Stable disease (SD) | 24
  Progressive disease (PD) | 4
  Not Evaluable (NE) | 21

2. Secondary Outcome: Kaplan-Meier Estimates of Progression Free Survival as Determined by the Independent Response Review Panel (IRRP)
Description: Progression-free survival was defined as the number of days from the date of first treatment to the date of first objective documentation of progressive disease (PD) as determined by the IRRP, or death due to any cause. Results are expressed in months.
  Progressive Disease (PD) was defined as an increase in size/number of nodes, size of liver or spleen, increase in lymphocytes, or aggressive histology.
Time Frame: up to 5 years
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alemtuzumab 30mg
Number analyzed (Participants) | 86
months | 12.43 [9.934 to 14.375]

3. Secondary Outcome: Kaplan-Meier Estimates of Duration of Response as Determined by the Independent Response Review Panel (IRRP)
Description: Duration of response was analyzed for participants who achieved a complete response (CR) or partial response (PR) and was defined as the number of days from the first date of documented response to the date of progressive disease (PD) as determined by IRRP or death due to any cause. Results are stated in months.
  Progressive Disease (PD) was defined as an increase in size/number of nodes, size of liver or spleen, increase in lymphocytes, or aggressive histology.
Time Frame: up to 5 years
Population: Participants who had a complete response or a partial response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alemtuzumab 30mg
Number analyzed (Participants) | 37
months | 11.09 [9.013 to 14.572]

4. Secondary Outcome: Kaplan-Meier Estimates of Overall Survival
Description: Overall survival was defined as the time in days from the date of first treatment to the date of death due to any cause for all participants. Results are stated in months.
Time Frame: up to 5 years
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alemtuzumab 30mg
Number analyzed (Participants) | 86
months | 38.29 [30.099 to NA] — values were not calculable since there were not enough events for the statistical estimation, ie, few participants died

5. Secondary Outcome: Participants With a Minimal Residual Disease (MRD) Status of Negative
Description: MRD negativity represents a very positive response outcome. MRD negativity in this report was defined by the absence of tumor cells in bone marrow, using 4-color flow cytometry. All patients are evaluated for treatment response based on National Cancer Institute Working Group (NCIWG) criteria. Of patients who have achieved a clinical complete response (CR) or partial response (PR) that met National Cancer Institute Working Group (NCIWG) criteria of CR except blood recovery, a bone marrow sample was taken for flow cytometry measure of MRD negativity.
Time Frame: 44 weeks
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Alemtuzumab 30mg
Number analyzed (Participants) | 86
participants | 4

6. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAE)
Description: Number of participants with treatment-emergent adverse events (TEAEs). AEs were graded by the investigator using the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 and were assessed for relatedness to study treatment (5 point scale from 'not related' to 'definitely related') and severity (5 point scale with grade 5 being most severe). Categories reported include participant counts for treatment-emergent AEs, injection site reactions, AEs for infections, serious AEs, AEs causing discontinuation of study drug(s), deaths and severity.
Time Frame: up to 18 weeks of treatment plus 45 days
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Alemtuzumab 30mg
Number analyzed (Participants) | 86
participants
  >=1 TEAE | 82
  >=1 TEAE related to drug | 80
  >=1 injection site reaction | 49
  >=1 injection site reaction related to drug | 48
  >=1 infection | 49
  >=1 infection related to drug | 35
  >=1 serious AE | 46
  >=1 serious AE related to drug | 39
  Discontinued study drug due to AE | 21
  Discontinued study drug due to related AE | 20
  Deaths | 12
  Deaths within 30 days of last dose | 3
  TEAE with worst severity grade 1 | 3
  TEAE with worst severity grade 2 | 8
  TEAE with worst severity grade 3 | 18
  TEAE with worst severity grade 4 | 45
  TEAE with worst severity grade 5 | 8

7. Primary Outcome: Percentage of Participants Who Had an Overall Response (OR) as Determined by the Independent Response Review Panel (IRRP)
Description: Participants were evaluated by the IRRP according to National Cancer Institute (NCI) 1996 response criteria. The percentage of participants whose best response observed during the study was either a Complete Response (CR) or a Partial Response (PR). Overall Response (OR) = CR + PR. A Complete Response (CR) exhibits a normal physical exam, marrow cells and blood values. A Partial Response (PR) has a >= 50% decrease from baseline in lymphocytes, lymphadenopathy and liver or spleen exam.
Time Frame: up to 44 weeks
Population: Full analysis set. 95% confidence interval calculated using exact binomial method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alemtuzumab 30mg
Number analyzed (Participants) | 86
percentage of participants | 43.0 [32.4 to 54.2]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs: up to 18 weeks of treatment plus 45 additional days
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables. Events are listed independent of relationship to treatment reported.
Arm/Group | Alemtuzumab 30mg
Serious Adverse Events (participants affected / at risk) | 46/86
Other Adverse Events (participants affected / at risk) | 81/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab 30mg (N=86)
Bone marrow failure (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Angina unstable (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Large intestine perforation (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chills (General disorders) | 2
Device dislocation (General disorders) | 1
Localised oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 6
Bile duct obstruction (Hepatobiliary disorders) | 1
Cholangitis acute (Hepatobiliary disorders) | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Abscess neck (Infections and infestations) | 1
Aspergillosis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Bronchopneumonia (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 3
Cytomegalovirus infection (Infections and infestations) | 9
Ear infection (Infections and infestations) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pneumonia fungal (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Fractured ischium (Injury, poisoning and procedural complications) | 1
Cytomegalovirus test positive (Investigations) | 2
Liver function test abnormal (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Polymyositis (Musculoskeletal and connective tissue disorders) | 1
Ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Richter's syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Encephalitis (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hypoglycaemic coma (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Oedema genital (Reproductive system and breast disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab 30mg (N=86)
Anaemia (Blood and lymphatic system disorders) | 28
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Haemolysis (Blood and lymphatic system disorders) | 2
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 27
Lymphopenia (Blood and lymphatic system disorders) | 14
Neutropenia (Blood and lymphatic system disorders) | 43
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 3
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 4
Ear pain (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Hypothyroidism (Endocrine disorders) | 1
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Erythema of eyelid (Eye disorders) | 1
Eye haemorrhage (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 5
Aphthous stomatitis (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 15
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Epigastric discomfort (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 17
Odynophagia (Gastrointestinal disorders) | 1
Peptic ulcer (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 3
Tongue coated (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 14
Asthenia (General disorders) | 6
Axillary pain (General disorders) | 1
Catheter site haematoma (General disorders) | 1
Chills (General disorders) | 20
Fatigue (General disorders) | 25
Hypothermia (General disorders) | 1
Influenza like illness (General disorders) | 1
Injection site erythema (General disorders) | 29
Injection site haematoma (General disorders) | 1
Injection site pain (General disorders) | 2
Injection site pruritus (General disorders) | 4
Injection site rash (General disorders) | 4
Injection site reaction (General disorders) | 14
Injection site swelling (General disorders) | 1
Malaise (General disorders) | 2
Oedema peripheral (General disorders) | 8
Pain (General disorders) | 6
Pyrexia (General disorders) | 30
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Drug hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Acute sinusitis (Infections and infestations) | 1
Balanitis candida (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 6
Escherichia urinary tract infection (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 7
Oesophageal candidiasis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oral fungal infection (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Oropharyngeal candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 4
Rhinitis (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 3
Sinusitis aspergillus (Infections and infestations) | 1
Systemic candida (Infections and infestations) | 1
Tinea capitis (Infections and infestations) | 1
Tinea infection (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 4
Arthropod bite (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 2
Thermal burn (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Beta 2 microglobulin increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Blood iron decreased (Investigations) | 1
Blood potassium decreased (Investigations) | 2
Blood pressure increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Body temperature increased (Investigations) | 1
CD4 lymphocytes decreased (Investigations) | 1
Cytomegalovirus test positive (Investigations) | 13
Eosinophil count increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Protein total decreased (Investigations) | 2
Serum ferritin increased (Investigations) | 1
Weight decreased (Investigations) | 8
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 12
Fluid retention (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3
Increased appetite (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Pseudohyperkalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Polymyositis (Musculoskeletal and connective tissue disorders) | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ageusia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 7
Dysarthria (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 16
Hemiparesis (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 4
Migraine (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 3
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 4
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 9
Mood altered (Psychiatric disorders) | 1
Neurosis (Psychiatric disorders) | 1
Stress (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Balanitis (Reproductive system and breast disorders) | 1
Breast oedema (Reproductive system and breast disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinusitis noninfective (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 9
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Night sweats (Skin and subcutaneous tissue disorders) | 12
Petechiae (Skin and subcutaneous tissue disorders) | 3
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 11
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 8
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 3
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 6
Orthostatic hypotension (Vascular disorders) | 3
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after an independent multi-investigator publication (in which the PI can participate) or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.